CLINICAL TRIAL: NCT04443712
Title: Screening for Patients Admitted to Ain-Shams University Hospitals for SARS-COV-2 (COVID19)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samia Girgis (Other)
Responsible Party: Sponsor-Investigator, Samia Girgis, vice director of ASU Hospitals, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: FMASU P29 /2020
Record Dates: First submitted 2020-06-16; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Disease 2019 (COVID19)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to screen the patients seeking hospitalization in Ain Shams university hospitals and identify a cost effective tool for continuing screening the patients all through the epidemic period

DETAILED DESCRIPTION:
Study setting: Ain-Shams University Hospitals. It is a campus including the following main hospitals: Gynecology and Obstetrics, Oncology, Pediatrics, Psychiatry, Internal Medicine, surgical, cardiothoracic and Geriatrics.

Study population: All patients needing admission in Ain-Shams University Hospitals are eligible for the study.

Sample size: There is no incidence data published till now. Only the confirmed detected cases have been reported. We assumed that the community cases are around 10 times that of detected cases.

it was estimated to be 1900 patients with 95% confidence level given the frequency of positive screening 0.05% with precision ± 0.1%. 10

The patients will be enrolled in the study using consecutive sample till the sample size is achieved.

Study methods:

Every enrolled patient will be subjected to:

1. An interview questionnaire including personal data ( age, gender, residence , contact details ) , epidemiological data (history of contact to a COVID-19 case, History of travel), clinical data history ( Fever, Cough, sore throat)
2. Reverse Transcription Polymerase Chain Reaction (RT-PCR)
3. Antibody IgM-IgG test for SARS-CoV-2

Statistical analysis:

Data will be validated, cleaned and entered in spreadsheet. SPSS program will be used for analysis.

Qualitative data will be presented in frequency and related percentage. Quantitative data with normal distribution will be presented in mean and standard deviation or median and interquartile for non-normally distributed data.

Incidence of positive screening test among the total will be calculated with 95% confidence interval.

Comparison between groups will be done using relevant suitable parametric or non-parametric tests. A "P" value of 0.05 is decided to be the level of significance.

Risk ratios will be calculated for estimation of risk with 95% confidence interval.

Cost per one positive detected screening test will be calculated (Total cost / total positive cases). The direct and indirect costs will be calculated by the laboratory department.

Ethical considerations:

The protocol will be submitted for approval by the University Ethical Research Committee.

The objectives and methods of the research will be explained to the participants.

An informed consent will be obtained from subjects willing to participate in the research and the subjects are free to withdraw from research anytime.

Confidentiality of the data will be highly secured. Positive cases will be reported to the Ministry of Health and Population (MOHP). The guidelines of isolation and treatment protocol of MOHP will be followed.

ELIGIBILITY:
Inclusion Criteria - All hospitalized patients in Ain-Shams University Hospitals.

Exclusion Criteria:

- Those who refuse to participate in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients needing admission in Ain-Shams University Hospitals; which is a campus including the following main hospitals: Gynecology and Obstetrics, Oncology, Pediatrics, Psychiatry, Internal Medicine, surgical, cardiothoracic and Geriatrics.
Sampling Method: Non-Probability Sample
Enrollment: 1900 (Estimated)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of the new COVID19 among hospitalized patients | 12 months
  To measure the incidence of the new SARS-COV-2 (COVID19) among patients seeking hospitalization to Ain-Shams University Hospitals

SECONDARY OUTCOMES:
Cost of screening hospitalized patients | 12 months
  To determine the cost of screening hospitalized patients

CONTACTS AND LOCATIONS:
Overall Officials: Samia Girgis, Principal Investigator — Vice Director of ASU Hospital
Locations (1):
- Faculty of Medicine Ain Shams University Research Institute- Clinical Research Center, Cairo, Non-US, Egypt

IPD SHARING:
Plan to Share IPD: No